CLINICAL TRIAL: NCT00358059
Title: Behavior Therapy for Families of Diabetic Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01DK043802 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2005-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes mellitus; adolescence; adherence; glycemic control; adaptation; communication
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Communication

INTERVENTIONS:
Behavioral: Behavioral Family Systems Therapy for Diabetes

SUMMARY:
Effective adaptation to type 1 diabetes mellitus requires adolescents and their families to work together effectively to solve problems and resolve disagreements in order to achieve acceptable diabetic control and treatment adherence. Many studies show that problematic family communication, insufficient parental involvement in care and parent-adolescent conflict are associated with poor adherence and poor diabetic control. This study tests a family communication and problem solving intervention by randomizing families of adolescent with type 1 diabetes to 6 months' treatment either with the experimental intervention, continuation in standard medical care for diabetes, or participation in a multifamily educational support group. Families are then followed for an additional 12 months to examine the longer-term effects of the interventions on the targeted diabetes outcomes.

DETAILED DESCRIPTION:
Adolescents with Type 1 diabetes mellitus often struggle to maintain adequate treatment adherence and diabetic control, leading to preventable hospitalizations and emergency room visits. Numerous cross-sectional and prospective studies show that family communication and conflict resolution skills are important influences on adolescents' diabetic control, treatment adherence and psychological adjustment. Empirical validation of psychological interventions targeting these processes could reduce excess health care costs and risks of diabetic complications. In the parent grant, we showed that Behavioral Family Systems Therapy (BFST; Robin & Foster, 1989) yielded improvements in family communication skills and parent-adolescent relationships, but it had weaker and less durable effects on treatment adherence and diabetic control. In this competing continuation application, we have relied on extensive preliminary data, our clinical experience with BFST and the results of others' investigations to formulate refinements to BFST that are designed to maximize its impact on diabetes treatment adherence and metabolic control. These include required targeting of behavioral barriers to adherence and diabetic control for every family, lengthening treatment from 3 to 6 months, and incorporation of several treatment components that were shown to be effective in other studies. We propose a randomized, controlled trial of this refined BFST intervention compared with standard medical therapy or participation in a diabetes educational support group on measures of: family communication, parent-adolescent relationships, adolescent psychological adjustment, treatment adherence, diabetic control and health care use. We will analyze predictors of treatment outcome and evaluate the clinical significance, social validity and maintenance of treatment effects over 6month and 12-month follow-up intervals. The results could influence the clinical practice of diabetes management and health care policy regarding adolescents with diabetes and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

Age of adolescent 12-<17 years Type 1 diabetes for >2 years Living in a home environment English reading ability at 5th grade level or above Established diabetes care at participating site Working telephone service Intent to remain living in same region for next 18 months -

Exclusion Criteria:

Presence of another chronic systemic disease Inpatient psychiatric treatment of patient or caregiver in prior 6 months Current outpatient treatment of psychosis, major depression or substance use disorder in parent/caregiver

-

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2000-10; Study Completion 2006-01

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c)
Treatment adherence

SECONDARY OUTCOMES:
Parent-adolescent communication
Family problem solving and conflict resolution skills
Diabetes-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wysocki, Ph.D., Principal Investigator — Nemours Children's Clinic
Locations (2):
- United States (2):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Washington University in St. Louis School of Medicine, St Louis, Missouri

REFERENCES:
- [Result] Wysocki T, Harris MA, Buckloh LM, Mertlich D, Lochrie AS, Taylor A, Sadler M, Mauras N, White NH. Effects of behavioral family systems therapy for diabetes on adolescents' family relationships, treatment adherence, and metabolic control. J Pediatr Psychol. 2006 Oct;31(9):928-38. doi: 10.1093/jpepsy/jsj098. Epub 2006 Jan 9. PMID 16401678